CLINICAL TRIAL: NCT00010088
Title: Study Of Gemcitabine, Leukovorin, And Fluorouracil Used To Treat Locally Advanced And Metastatic Pancreatic And Biliary Adenocarcinomas
Brief Title: Chemotherapy in Treating Patients With Locally Advanced or Metastatic Cancer of the Pancreas or Bile Duct
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068440; FRE-GERCOR-FOLFUGEM2-D99-3; EU-20024
Record Dates: First submitted 2001-02-02; First posted 2004-05-20 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2007-04

CONDITIONS: Extrahepatic Bile Duct Cancer; Pancreatic Cancer
Keywords: stage II pancreatic cancer; stage III pancreatic cancer; unresectable extrahepatic bile duct cancer; adenocarcinoma of the extrahepatic bile duct; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Pancreatic Neoplasms | interventions — Fluorouracil; Gemcitabine; Leucovorin; Radiotherapy

INTERVENTIONS:
Drug: fluorouracil
Drug: gemcitabine hydrochloride
Drug: leucovorin calcium
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining gemcitabine, leucovorin, and fluorouracil in treating patients who have locally advanced or metastatic cancer of the pancreas or bile duct.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate, in terms of WHO objectives and clinical benefit, in patients with locally advanced or metastatic pancreatic or biliary adenocarcinoma treated with gemcitabine, leucovorin calcium, and fluorouracil. II. Determine the tolerance of this regimen in this patient population. III. Determine the survival without disease progression in patients treated with this regimen. IV. Determine the overall survival in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients receive leucovorin calcium IV over 2 hours followed by fluorouracil IV over 24 hours on day 1 followed by gemcitabine IV over 80-150 minutes on day 2. Treatment repeats every 2 weeks for a minimum of 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving complete response may continue chemotherapy for up to 1 year. Patients with locally advanced disease after 3 months of chemotherapy may receive concurrent radiotherapy with chemotherapy for 5 weeks, or may undergo surgical resection. Fluorouracil-based chemotherapy (with or without radiotherapy) may then resume after surgery. Patients are followed for survival.

PROJECTED ACCRUAL: A total of 14-39 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed pancreatic or biliary duct adenocarcinoma Metastatic or locally advanced No cerebral metastasis Surgically unresectable

PATIENT CHARACTERISTICS: Age: 18 to 75 Performance status: ECOG 0-2 Life expectancy: More than 12 months Hematopoietic: Absolute neutrophil count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Alkaline phosphatase less than 5 times normal Bilirubin less than 1.5 times normal Renal: Creatinine less than 1.5 times normal No uncontrolled or persistent hypercalcemia Cardiovascular: No severe cardiac failure Pulmonary: No severe respiratory failure Other: No other malignant tumor considered incurable or untreatable No uncontrolled pain No psychological, familial, social, or geographical reasons that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: No concurrent corticosteroids except as antiemetic Radiotherapy: No prior radiotherapy Surgery: See Disease Characteristics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-01

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Louvet, MD, PhD, Study Chair — Hopital Saint Antoine
Locations (50):
- France (49):
  - Clinique De Rochebelle, Alès
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Centre D'Oncologie Du Pays-Basqu, Bayonne
  - C.H.G. Beauvais, Beauvais
  - Institut Bergonie, Bordeaux
  - CMC Bligny, Briis-sous-Forges
  - Clinique Saint-Jean, Cagne-sur-Mer
  - Hopital Fontenoy, Chartres
  - Hopital Beaujon, Clichy
  - Hopital Drevon, Dijon
  - Centre D'Oncologie Dunkerquois, Dunkirk
  - Polyclinique De La Foret, Fontaineblea
  - CHR de Grenoble - La Tronche, Grenoble
  - Centre De Charlebourg, La Garenne-Colombes
  - Clinique Du Cap D'OR, LA Seyne Sur Me
  - Hopital Andre Mignot, Le Chesnay
  - Hopital de la Croix Rousse, Lyon
  - Assistance Publique Hopitaux de Marseille Hopitaux Sud, Marseille
  - Hopital Notre-Dame de Bon Secours, Metz
  - Hopital Clinique Claude Bernard, Metz
  - Intercommunal Hospital, Montfermeil
  - Centre Hospitalier De Moulins Yzeure, Moulins
  - Centre Hospitalier de Mulhouse, Mulhouse
  - CHR Hotel Dieu, Nantes
  - American Hospital of Paris, Neuilly-sur-Seine
  - CHR D'Orleans - Hopital de la Source, Orléans
  - Hopital Laennec, Paris
  - Clinique Du Mont Louis, Paris
  - Hopital Rothschild, Paris
  - Hopital Saint Joseph, Paris
  - L'Institut Mutualiste Montsouris Jourdan, Paris
  - Hopital Boucicaut, Paris
  - Hopital Saint-Louis, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Tenon, Paris
  - Hopital De La Croix, Paris
  - Clinique Bizet, Paris
  - Hopital Haut Leveque, Pessac
  - Clinique Ste-Marie, Pontoise
  - Hopital Claude Gallien, Quincy-sous-Sénart
  - Polyclinique De Courlancy, Reims
  - Oncologie Medicale, Saint-Jean
  - Centre du Rouget, Sarcelles
  - C.H. Senlis, Senlis
  - Centre Hospitalier Intercommunal Toulon - La Seyne/Mer, Toulon
  - Clinique Pasteur, Toulouse
  - Polyclinique Flemming, Tours
  - Centre Saint-Yves, Vannes
  - Institut Gustave Roussy, Villejuif
- Hopital de la Ville D'Esch-sur-Alzette, Esch-sur-Alzette, Luxembourg

REFERENCES:
- [Background] Huguet F, Andre T, Hammel P, Artru P, Balosso J, Selle F, Deniaud-Alexandre E, Ruszniewski P, Touboul E, Labianca R, de Gramont A, Louvet C. Impact of chemoradiotherapy after disease control with chemotherapy in locally advanced pancreatic adenocarcinoma in GERCOR phase II and III studies. J Clin Oncol. 2007 Jan 20;25(3):326-31. doi: 10.1200/JCO.2006.07.5663. PMID 17235048
- [Result] Andre T, Noirclerc M, Hammel P, Meckenstock R, Landi B, Cattan S, Selle F, Codoul JF, Guerrier-Parmentier B, Mokhtar R, Louvet C; GERCOR. Phase II study of leucovorin, 5-fluorouracil and gemcitabine for locally advanced and metastatic pancreatic cancer (FOLFUGEM 2). Gastroenterol Clin Biol. 2004 Aug-Sep;28(8-9):645-50. doi: 10.1016/s0399-8320(04)95042-7. PMID 15646530